CLINICAL TRIAL: NCT00638300
Title: Removal of Ligand-bound Iron During Intravenous Iron Administration in Hemodialysis by Large Pore Dialyzers
Brief Title: Removal of Ligand-bound Iron During Intravenous (IV) Iron Administration in Hemodialysis (HD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Collaborators: Bnai Zion Medical Center (Other Government); Rivka Ziv Medical Center (Unknown)
Responsible Party: David Tovbin MD, Soroka University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: sor421306ctil
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2008-03

CONDITIONS: Hemodialysis Patients
Keywords: hemodialysis; iron; inflammation; atomic absorption; dialysate; advanced oxidation protein products; large pore dialysate; bicarbonate; calcium; citrate; ligand
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): large pore dialyzers (FX80, Fresenius, Germany)
  Interventions: Device: large pore (FX80) compared to small pore dialyzer (F8HPS)
- 2 (Experimental): small pore dialyzers ( F8HPS, Fresenius, Germany)
  Interventions: Device: large pore (FX80) compared to small pore dialyzer (F8HPS)
- A (Experimental): dialysate bicarbonate concentration of 33 mEq/l
  Interventions: Other: Dialysate bicarbonate of 33 mEq/L compared to 40 mEq/L
- B (Experimental): dialysate bicarbonate concentration of 40 mEq/l
  Interventions: Other: Dialysate bicarbonate of 33 mEq/L compared to 40 mEq/L
- I (Experimental): dialysate calcium concentration of 3 mEq/L
  Interventions: Other: Dialysate calcium of 3 mEq/L compared to 2.5 mEq/L
- II (Experimental): dialysate calcium concentration of 2.5 mEq/L
  Interventions: Other: Dialysate calcium of 3 mEq/L compared to 2.5 mEq/L

INTERVENTIONS:
Device: large pore (FX80) compared to small pore dialyzer (F8HPS) — Effect of pore size
  Arms: 1; 2
Other: Dialysate bicarbonate of 33 mEq/L compared to 40 mEq/L — Effect of dialysate bicarbonate concentration
  Arms: A; B
Other: Dialysate calcium of 3 mEq/L compared to 2.5 mEq/L — Effect of dialysate calcium concentration
  Arms: I; II

SUMMARY:
The study's hypothesis is that HD with large pore dialyzers remove to the dialysate iron which is bound to potentially dialyzable ligands, after it's release from intravenous iron compound administered during hemodialysis.

DETAILED DESCRIPTION:
Most hemodialysis(HD) patients receive during HD intravenous iron compounds, which are composed of an iron core and a sugar polymer shell.

A small percentage of iron from the iron compound is released to the plasma, and may be associated with increased oxidative stress and protein oxidation. The study's hypothesis is that HD with large pore dialyzers may remove to the dialysate iron which is bound to potentially dialyzable ligands, after it's release from intravenous iron compound administered during hemodialysis.

Ligand-bound iron removal is also hypothesized to be affected by dialysate calcium and bicarbonate concentrations, which may affect iron-ligand binding.

Study Specific aims are:

To evaluate

1. Iron removal assessing dialysate iron levels.
2. Effect of iron removal and it's associated experimental conditions on patient status, assessing plasma AOPP levels and inflammation related parameters

Study include 3 parts

1. Comparing large to small pore dialyzers

   (To achieve baseline uniform conditions, patients will be on uniform dialysate bicarbonate and calcium concentrations of 33 mEq/L and 3 mEq/L,respectively, using large pore dialyzers during this part, besides the 2 HD sessions evaluating low pore dialyzers)

   and after few week break

   Using large pore dialyzers to compare
2. Low to high dialysate bicarbonate concentration (using uniform dialysate calcium concentrations of 3 mEq/L)

   and after few week break
3. Low to high dialysate calcium concentrations concentration (using uniform dialysate bicarbonate of 33 mEq/L)

In each part, patients will be first evaluated in HD without IV iron administration, which will serve as a control for evaluation after a week in HD with IV iron administration.

In each part, patients will be randomized to start either with one of the 2 experimental conditions, and after 1 week without evaluation will cross-over to the other experimental condition.

Patients may participate in 1,2 or the 3 parts of study depending on their will and condition.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients

Exclusion Criteria:

* Acute disease (infection, thrombosis, ischemia, bleeding) Hepatitis B, Hepatitis C or HIV
* Intravenous iron administration or packed red cell transfusion in the last 3 weeks prior to the study
* Refusal to comply with limitations in fat containing food during HD with plasma sampling for AOPP evaluation

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
1. Dialysate Iron levels 2. Plasma levels of advanced oxidation protein products(AOPP) | Before HD, after 1 hour of HD with or without IV iron and at end of HD

CONTACTS AND LOCATIONS:
Overall Officials: David Tovbin, MD, Principal Investigator — Soroka University Medical Center
Locations (3):
- Israel (3):
  - HD unit in Department of Nephrology in Soroka Universty Medical Center, Beersheba
  - HD unit in Bnai-zion Medical Center, Haifa
  - Rivka Ziv Medical center, Safed